CLINICAL TRIAL: NCT05649722
Title: An Open-Label Extension Study to Assess the Safety, Tolerability, and Effectiveness of the Long-Term Use of Treprostinil Palmitil Inhalation Powder in Participants With Pulmonary Hypertension Associated With Interstitial Lung Disease
Brief Title: An Extension Study of Treprostinil Palmitil Inhalation Powder (TPIP) for Pulmonary Hypertension Associated With Interstitial Lung Disease (PH-ILD)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INS1009-212; 2022-001950-45 (EudraCT Number); 2023-505540-19-00 (Other: EU CT Number)
Expanded Access: NCT06939647 (Available)
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Hypertension; Interstitial Lung Disease
Keywords: Treprostinil Palmitil
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treprostinil Palmitil Inhalation Powder (Experimental): Participants who are not transitioning immediately from INS1009-211 and other lead-in studies, will be administered TPIP, once daily (QD), during 3-week titration period.
  Participants who are transitioning immediately from a randomized blinded lead-in TPIP study and who previously received:
  1. TPIP- will be administered placebo QD along with the maximum tolerated dose (MTS) TPIP dose from lead-in study in a blinded manner during 3-week titration period.
  2. Placebo- will be administered TPIP QD along with the achieved placebo dose from lead-in study in a blinded manner during 3-week titration period.
  The overall treatment period will be 24 months.
  Interventions: Drug: Treprostinil Palmitil Inhalation Powder; Drug: Placebo

INTERVENTIONS:
Drug: Treprostinil Palmitil Inhalation Powder — Oral inhalation using a capsule-based dry powder inhaler device.
  Other Names: INS1009
Drug: Placebo — Oral placebo inhalation using a capsule-based dry powder inhaler device.

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of the long-term use of TPIP in participants with PH-ILD from Study INS1009-211 (NCT05176951) and other lead-in studies of TPIP in participants with PH-ILD.

ELIGIBILITY:
Inclusion Criteria:

* Participants who completed the end of treatment visit in Study INS1009-211 (NCT05176951). Participants for whom the OLE study was not available at the time of their completion of the lead-in study are eligible for enrolment within one year of their lead-in end of treatment visit.
* Complete baseline screening assessments to confirm eligibility to participate if more than 30 days have elapsed since the end of the study visit in Study INS1009-211, or any other lead-in PH-ILD TPIP study.
* Capable of giving signed informed consent that includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Participants who experienced any hypersensitivity or adverse drug reaction or were withdrawn early/discontinued in a previous PH-ILD TPIP study, which in the opinion of the Investigator, could indicate that continued treatment with TPIP may present an unreasonable risk for the participant.
* Initiation of parenteral administration of prostacyclin analogues (eg, TRE, epoprostenol) since the completion of Study INS1009-211 or other TPIP studies. Initiation of inhaled prostacyclin analogues (eg, TRE [Tyvaso] or iloprost) and oral prostacyclin analogues (eg, TRE [Orenitram]) or receptor agonists (eg, selexipag) are permitted if stopped 24 hours prior to the start of study drug administration.

Pregnant or breastfeeding. Male and female participants must use contraceptives that are consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Female participants of childbearing potential must have a negative urine pregnancy test result at trial entry before the first dose of study drug.

- Any medical or psychological condition, including relevant laboratory abnormalities at screening that, in the opinion of the Investigator, suggest a new and/or insufficiently understood disease that may present an unreasonable risk to the study participant as a result of participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experienced a Treatment Emergent Adverse Event (TEAE) | Up to approximately 25 months

SECONDARY OUTCOMES:
Absolute Change From Pre-Open-Label Extension (OLE) Baseline in 6-Minute Walk Distance (6MWD) | Pre-OLE Baseline (Baseline of the lead-in TPIP study) to Months 6, 12, 18, and 24
Relative Change From Pre-OLE Baseline in 6-MWD | Pre-OLE Baseline (Baseline of the lead-in TPIP study) to Months 6, 12, 18, and 24
Change From Pre-OLE Baseline in Forced Vital Capacity (FVC) | Pre-OLE Baseline (Baseline of the lead-in TPIP study) to Months 6, 12, 18, and 24
Change From Pre-OLE Baseline in Percent Predicted FVC (FVC%) | Pre-OLE Baseline (Baseline of the lead-in TPIP study) to Months 6, 12, 18, and 24
Change From Pre-OLE Baseline in Forced Expiratory Volume in 1 Second (FEV1) | Pre-OLE Baseline (Baseline of the lead-in TPIP study) to Months 6, 12, 18, and 24
Change From Pre-OLE Baseline in Percent Predicted FEV1 (FEV1%) | Pre-OLE Baseline (Baseline of the lead-in TPIP study) to Months 6, 12, 18, and 24
Change From Pre-OLE Baseline in Forced Expiratory Flow Between 25% and 75% of Forced Vital Capacity (FEF25-75%) | Pre-OLE Baseline (Baseline of the lead-in TPIP study) to Months 6, 12, 18, and 24
Absolute Change From Pre-OLE Baseline in Lung Diffusion Capacity for Carbon Monoxide (DLCO) | Pre-OLE Baseline (Baseline of the lead-in TPIP study) to Months 12 and 24
Relative Change From Pre-OLE Baseline in Lung DLCO | Pre-OLE Baseline (Baseline of the lead-in TPIP study) to Months 12 and 24
Change From Pre-OLE Baseline in the Concentration of N-Terminal Fragment B-Type Natriuretic Peptide (NT-proBNP) in Blood | Pre-OLE Baseline (Baseline of the lead-in TPIP study) to Months 6, 12, 18, and 24
Annualized Rate of Clinical Worsening Events Based on Percentage of Participants With Clinical Worsening Events | Up to Month 24
  Clinical worsening events are defined as one of the following: Hospitalization due to a cardiopulmonary indication; Lung transplantation; Death from any cause; Decrease in 6MWD ≥ 15% from baseline; Directly related to disease under study, at 2 consecutive visits at least 24 hours apart; Need for additional pulmonary hypertension (PH) therapy. Annualized clinical worsening event rate is defined as the total number of clinical worsening events that occurred during the treatment period divided by the total number of participant-years during the treatment period.
Annualized Rate of Occurrence of Acute Exacerbations of Underlying Interstitial Lung Disease (AE-ILDs) | Up to Month 24
Change From OLE Baseline in the King's Brief Interstitial Lung Disease (K-BILD) Questionnaire Score | OLE Baseline (Day 1) to Months 6, 12, 18, and 24
Change From OLE Baseline in the Euro Quality of Life-5 Dimension-5 Level (EQ-5D-5L) Questionnaire Score | OLE Baseline (Day 1) to Months 6, 12, 18, and 24
Plasma Concentration Levels of Treprostinil Palmitil (TP) and Treprostinil (TRE) | OLE Baseline (Day 1), Months 6, 12, 18, and 24

CONTACTS AND LOCATIONS:
Locations (22):
- Argentina (2):
  - ARG003, Autonomus City of Buenos Aires, Buenos Aires
  - ARG001, Rosario, Santa Fe Province
- AUS005, Macquarie Park, New South Wales, Australia
- BEL002, Liège, Belgium
- Germany (7):
  - GER006, Heidelberg, Baden-Wurttemberg
  - GER004, München, Bavaria
  - GER010, Giessen, Hesse
  - GER003, Essen, North Rhine-Westphalia
  - GER001, Dresden, Saxony
  - GER002, Berlin
  - GER012, Berlin
- Italy (4):
  - ITA004, Milan, Lombardy
  - ITA002, Monza, Lombardy
  - ITA001, Palermo, Sicily
  - ITA003, Napoli
- Spain (5):
  - ESP003, Palma, Balearic Islands
  - ESP009, Santiago de Compostela, Galicia
  - ESP007, Oviedo, Principality of Asturias
  - ESP005, Barcelona
  - ESP010, Barcelona
- United Kingdom (2):
  - GBR003, Clydebank, Glasgow
  - GBR001, Sheffield, South Yorkshire

IPD SHARING:
Plan to Share IPD: No